CLINICAL TRIAL: NCT02617225
Title: Evaluation of DHaAL Intervention of Group Handwashing With Soap Before Mid-day Meals in Rural Elementary School of Assam
Brief Title: Effect of a Pilot Group Hand-washing Program on Handwashing Behaviors Among Elementary School Children in Assam
Status: Completed | Type: Observational
Sponsor: Network for Engineering and Economics Research and Management (Other)
Collaborators: UNICEF (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/06/UNICEF01
Record Dates: First submitted 2015-11-27; First posted 2015-11-30 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Handwashing Behaviors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- DHaAL Intervention: The group receives standard Ailment-free Life (DHaAL) DHaAL intervention
  Interventions: Behavioral: DHaAL Intervention
- DHaAL +CFSS Intervention: This group received the standard DHaAL intervention and additional support under another UNICEF program named Child Friendly School System (CFSS).
  Interventions: Behavioral: DHaAL Intervention; Behavioral: DHaAL + CFSS Intervention
- Control: This group receive the standard / business-as-usual support from the Education Department, but does not receive DHaAL or CFSS Interventions.

INTERVENTIONS:
Behavioral: DHaAL Intervention — This group handwashing program is for rural elementary schools to institutionalize the practice of handwashing before mid-day meal consumption and after use of toilets by harnessing the theory of social peer pressure.
  DHaAL intervention consists of: (1) capacity building of school teachers to implement group handwashing; (2) installing group handwashing station; (3) generating demand among students to wash hands in group; and (4) establishing systems to sustain handwashing infrastructure and behaviors.
  Groups: DHaAL +CFSS Intervention; DHaAL Intervention
Behavioral: DHaAL + CFSS Intervention — In addition to support under DHaAL, several intervention schools receive a more holistic and participatory support that focuses on health, safety, nutrition status, and psychological wellbeing of the children, and thus can also influence handwashing practices (and other WASH facilities). CFSS provides capacity building support and establishes systems to improve school environment, learning outcome, teachers capacity, and physical education for children.
  Groups: DHaAL +CFSS Intervention

SUMMARY:
The United Nation's International Children's Emergency Fund (UNICEF) is supporting Saba Shikha Abihyan (SSA) (Education-for-All Mission) of the Government of Assam (GoA) under their Water-Sanitation-Hygiene in School (WinS) program to improve WASH facilities, practices and institutionalize WASH in school settings. Under the WinS program, UNICEF piloted a group hand washing program in 100 elementary schools. Multiple past studies have shown that handwashing is an effective intervention to reduce diarrheal diseases and respiratory tract infections, but the evidence on the interventions or programs that can achieve this behavior change is mixed and limited in case of school setting. The main objective of Daily Handwashing for an Ailment-free Life (DHaAL) program was to institutionalize handwashing with soap before consuming mid-day meals and after using toilets among elementary school students. DHaAL is implemented on the Mid-day Meal platform where free meals are given to all students attending government schools.

In addition to the standard DHaAL intervention, several pilot phase schools also received an additional program for a holistic and participatory development of school systems for health, nutrition, learning outcomes and wellbeing of children called Child Friendly School System (CFSS). Although CFSS is not a WASH intervention it can develop systems and processes and offer longer support from and implementing agencies which help DHaAL Intervention also.

This evaluation study seeks to answer whether DHaAL improved handwashing practice before the mid-day meals in rural lower primary schools as a primary research question. The intermediate outputs and secondary outcomes evaluated in this study include functionality of handwashing infrastructure at school, handwashing practice after toilet use, and availability of and use of handwashing facilities at homes (indirect effect). The evaluation study has other supplemental operations research objectives to help improve the program in future.

ELIGIBILITY:
Inclusion Criteria:

* Should be present in the school on the day of interview/survey

Exclusion Criteria:

* None

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Elementary schools (Class 1-5) from five education blocks in Kamrup district. The respondents/participants include school teachers (Interview/observations), Class 1-5 students (distant observation), Class 3-5 students (personal Interviews/observations) and their parents/other household members (personal Interview/observations).
Sampling Method: Probability Sample
Enrollment: 823 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of Class 1-5 children washing hands with soap before consuming mid-day meals in schools | On the day of interview (~12-24 months after the external support under DHaAL ceased)

SECONDARY OUTCOMES:
Proportion of Class 1-5 children washing hands with soap after the use of toilets for defecation or urination in schools | On the day of interview (~12-24 months after the external support under DHaAL ceased)
Proportion of schools having a functional handwashing station with water and soap | On the day of interview (~12-24 months after the external support under DHaAL ceased)
Proportion of households having a functional handwashing station with water and soap | On the day of interview (~12-24 months after the external support under DHaAL ceased)
  This is an indirect or spill over effect of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Patil, Principal Investigator — Network for Engineering and Economics Research and Management
Locations (1):
- NEERMAN, Mumbai, Maharashtra, India